CLINICAL TRIAL: NCT03260985
Title: Precision Psychiatry Continuity Clinic Project
Acronym: PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Leanne Williams, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 41868
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorders; Depressive Symptoms; Anxiety Disorders and Symptoms; Psychological Distress; Mood Disorders
MeSH Terms: conditions — Depressive Disorder; Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback Group (Experimental): All participants in the study will undergo a comprehensive neuroscience assessment including clinical questionnaires, a structured diagnostic interview, neuropsychological assessment, genetic testing, and structural and functional MRI. Participants randomized to the Feedback Group will have the results of this assessment shared with their psychiatric treatment team before they begin treatment. This data will be used at the full discretion of the treatment team to inform personalized treatment options. All treatment decisions remain up to the treatment providers and patient.
  Interventions: Other: Feedback Report
- Delayed Feedback Group (No Intervention): All participants in the study will undergo a comprehensive neuroscience assessment including clinical questionnaires, a structured diagnostic interview, neuropsychological assessment, genetic testing, and structural and functional MRI. However, participants randomized to the Delayed Feedback Group will not have the results of this assessment shared with their treatment team until the end of their participation in this study (12 weeks).

INTERVENTIONS:
Other: Feedback Report — A report of the data from the comprehensive neuroscience assessment is provided to the patient's care team.
  Arms: Feedback Group

SUMMARY:
This is a demonstration project focused on translating neuroscience insights into clinical practice. The researchers will evaluate how neuroscience assessments may be applied in the clinical setting to help inform care decisions. The aim of the study is to undertake a pragmatic pilot trial to assess whether the inclusion of structured feedback from neuroscience assessments has an effect on improving patient outcomes. The study will investigate how neuroscience assessments can be integrated into and improve clinical care. The impact of sharing information and conclusions from these assessments with psychiatric providers will be explored. Outcomes will include symptoms, social/occupational function and qualify of life.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Fluent and literate in English, and able to understand task instructions
* fMRI scanning eligibility, including no evidence of any form of metal embedded in the body (e.g., metal wires, nuts, bolts, screws, plates, sutures)
* Must be referred for treatment at the Stanford Department of Psychiatry Continuity Clinic

Exclusion Criteria:

* Presence of suicidal ideations representing imminent risk
* General medical condition, disease or neurological disorder that interferes with the assessments
* Traumatic brain injury (history of physical brain injury or blow to the head resulting in loss of consciousness greater than five minutes) and which could interfere with doing the assessments
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with ability to complete the assessments, or are unable and/or unlikely to follow the study protocols
* Pregnancy
* Presence of acute psychosis, schizophrenia spectrum, or other psychotic disorders
* Concurrent participation in intervention or treatment studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 weeks
  A 9-item questionnaire of self-reported symptoms of major depression commonly used in research and routine clinical care
Generalized Anxiety Disorder Questionnaire (GAD-7) | 12 weeks
  A 7-item questionnaire of self-reported symptoms of generalized anxiety commonly used in research and routine clinical care

SECONDARY OUTCOMES:
Sheehan Disability Scale (SDS) of Social/Occupational Functioning | 12 weeks
  Level of functioning in social, occupational, and home life domains
Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER) | 12 weeks
  Burden of side effects from psychiatric medication

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Williams, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Center for Cognitive and Neurobiological Imaging (CNI), Stanford, California, United States